CLINICAL TRIAL: NCT05673226
Title: Organosilane for Surface Cleaning in Intensive Care Units: A Cluster Randomized, Controlled, Crossover, Clinical Trial
Brief Title: Organosilane for Surface Cleaning in Intensive Care Units
Acronym: ORG-CLEAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Hospital Sirio-Libanes (Other); Hospital Moinhos de Vento (Other); Hospital Alemão Oswaldo Cruz (Other); Hospital do Coracao (Other); Beneficência Portuguesa de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 52639521.1.1001.0071
Record Dates: First submitted 2022-12-07; First posted 2023-01-06 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2023-11

CONDITIONS: Infection, Hospital
Keywords: Infection Control; Infections; Intensive Care Units; Pneumonia, Ventilator Associated; Catheter-Related Infections; Urinary Tract Infections; Organosilanes; Costs and Cost Analyses
MeSH Terms: conditions — Cross Infection; Infections; Pneumonia, Ventilator-Associated; Catheter-Related Infections; Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, cluster, crossover, trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surface disinfection with organosilane (Experimental): Organosilane will be sprayed on the surfaces, using an atomizer. When the environment has been completely covered (i.e., when all surfaces and equipment have a slightly damp film), we will proceed with the second phase of the disinfection of all heavily touched surfaces. surfaces of the bed, with a microfiber cloth with organosilane.
  Interventions: Other: Surface disinfection with Organosilane
- Usual surface disinfection (No Intervention): The control group will perform standard cleaning and disinfection of the beds and the environment according to their previous protocols, using the usual products.

INTERVENTIONS:
Other: Surface disinfection with Organosilane — Organosilane will be sprayed on the surfaces, using an atomizer. When the environment has been completely covered (i.e., when all surfaces and equipment have a slightly damp film), we will proceed with the second phase of the disinfection of all heavily touched surfaces. surfaces of the bed, with a microfiber cloth with organosilane.
  Arms: Surface disinfection with organosilane

SUMMARY:
The purpose of this study is to evaluate if surface disinfection with organosilane associated with traditional cleaning reduces the incidence of healthcare-associated infections (HAIs) in intensive care units when compared with traditional cleaning alone.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 years and older who will be admitted to the participating ICUs

Exclusion Criteria:

* Patients under 18 years
* ICUs that may use any organosilane formulation for surface disinfection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10301 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Incidence of healthcare associated infections | 6 months

SECONDARY OUTCOMES:
Contamination of environmental surfaces by multi-resistant microorganisms | 6 months
  We will collect environmental samples from 4 surfaces highly touched by the patient, health team and family (bed rails, monitor and infusion pump buttons, meal table or procedure table, and IV drip stand) before and after the intervention. (end of the 6 months). For analysis of the environmental samples, characterization of the density and microbiological profile of biofilms on the different surfaces of the ICU beds will be performed using large-scale DNA sequencing techniques associated with bioinformatics analysis.
Incidence of ventilator-associated pneumonia | 6 months
Incidence of central line-associated blood stream infections | 6 months
Incidence of catheter-associated urinary tract infection | 6 months
Intensive care unit length of stay costs | 6 months

CONTACTS AND LOCATIONS:
Locations (14):
- Brazil (14):
  - Hospital Jean Bittar, Belém
  - Santa Casa de Misericórdia, Belo Horizonte
  - Hospital de Base do Distrito Federal, Brasília
  - Hospital Universitário de Brasília, Brasília
  - Hospital Otoclínica, Fortaleza
  - Hospital Geral de Goiânia, Goiânia
  - Hospital do Tricentenário, Olinda
  - Hospital Escola Universidade Federal de Pelotas, Pelotas
  - Hospital Ernesto Dornelles, Porto Alegre
  - Hospital Ana Nery, Salvador
  - Hospital Santa Cruz, Santa Cruz do Sul
  - Hospital Presidente Vargas, São Luís
  - A.C. Camargo Cancer Center, São Paulo
  - Hospital do Coração, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, Analytic Code